CLINICAL TRIAL: NCT07125989
Title: Effect of Exercise Ventilatory Support Pressure on Endurance in Patients With Severe Chronic Obstructive Pulmonary Disease - AVE-BPCO
Acronym: AVE-BPCO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 24CH126; 2025-A00555-44 (Other: ANSM)
Record Dates: First submitted 2025-08-04; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic obstructive pulmonary disease; respiratory rehabilitation; non-invasive ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low intensity (Sham Comparator): Non-invasive ventilation less han 6 cmH2O
  Interventions: Device: non-invasive ventilation
- Moderate intensity (Active Comparator): Non-invasive ventilation 13 +/-3 cmH2O
  Interventions: Device: non-invasive ventilation
- High intensity (Experimental): Non-invasive ventilation 21 +/-3 cmH2O
  Interventions: Device: non-invasive ventilation

INTERVENTIONS:
Device: non-invasive ventilation — During the patient's first three respiratory rehabilitation sessions, each test on the cycle ergometer will be performed at 70% of maximum power (defined during the initial oxygen consumption (VO2) test) with ventilatory assistance at a different intensity (Low, moderate or high intensity).

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a chronic respiratory disease characterized by progressive obstruction of the airways. In advanced stages, it can progress to chronic respiratory failure with major respiratory repercussions.

Biologically, hyperinflation manifests as alveolar hypoventilation, which causes hypercapnia. Mechanically, it is responsible for an increase in ventilatory work associated with diaphragmatic muscle dysfunction and fatigue, leading to exercise incapacity.

Physical inactivity is a major predictor of mortality in patients with COPD. The recommendations of the European Respiratory Society (ERS) and the American Thoracic Society (ATS) emphasize the importance of exercise in the treatment and management of COPD.

Respiratory rehabilitation has been shown to have an indisputable effect on dyspnea and the quality of life of COPD patients. Current guidelines for respiratory rehabilitation recommend interventions at a frequency of at least 2 to 3 supervised high-intensity training sessions per week. A minimum of 4 weeks of physical training is necessary to achieve a significant improvement in quality of life, dyspnea, and endurance.

A reduction in the duration and intensity of sessions is often necessary, thus limiting the desired benefits of respiratory rehabilitation.

Non-invasive ventilation (NIV) provides mechanical respiratory assistance by helping inspiration and optimizing expiration through a non-invasive interface such as a mask. Its use during exercise in severe COPD is to try to correct hypercapnia, reduce dynamic hyperinflation by helping the respiratory muscles to improve their work, and reduce dyspnea and the feeling of muscle weakness.

However, the modalities in terms of ventilation mode and inspiratory support pressures are not clearly established.

DETAILED DESCRIPTION:
The objective of this study is therefore to compare different levels of ventilatory assistance during exercise to determine whether the level of inspiratory assistance during exercise significantly improves endurance in these patients and, in particular, whether high-intensity ventilatory assistance (inspiratory assistance 21 +/- 3 cmH20) provides a greater benefit in terms of endurance time compared to moderate intensity (inspiratory assistance 13 +/- 3 cmH20) or low intensity (inspiratory assistance < 6 cmH20).

ELIGIBILITY:
Inclusion Criteria:

* -COPD stage GOLD III or IV
* Baseline hypercapnia PaCO2 > 45 mmHg OR Alveolar hypoventilation during exercise (increase in PaCO2 > 5 mmHg),
* Exhaustion of more than 80% of ventilatory reserve OR max power < 50 Watts
* Affiliation or entitlement to social security coverage
* Signature of informed consent

Exclusion Criteria:

* BMI > 35
* Recent acute respiratory exacerbation < 4 weeks
* Severe unstable cardiac disease
* Pneumothorax or pneumomediastinum
* Pathological hypotension
* Cerebrospinal fluid leak, recent head trauma, or cranial surgery
* Severe bulbar disorder
* Dehydration
* Severe orthopedic or neurological disorder compromising rehabilitation.
* Patient deprived of liberty or patient under guardianship
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Pedaling time limit (in seconds) | Day 1, Day 3, Day 5
  Endurance capacity will be measured by the time limit for pedaling (in seconds) on a cycloergometer, performed during a respiratory rehabilitation session, at 70% of the maximum power developed during the maximum test.

SECONDARY OUTCOMES:
Partial pressure of oxygen (PaO2) in mmHg | Day 1, Day 3, Day 5
  PaO2 measured by capillary blood gas analysis performed at peak exercise during a respiratory rehabilitation session
Partial pressure of carbon dioxide (PaCO2) in mmHg | Day 1, Day 3, Day 5
  PaCO2 measured by capillary blood gas analysis performed at peak exercise during a respiratory rehabilitation session
Lactate in mmol/l | Day 1, Day 3, Day 5
  Lactate measured by capillary blood gas analysis performed at peak exercise during a respiratory rehabilitation session
Peripheral muscle oxygenation (% SmO2) | Day 1, Day 3, Day 5
  Measurement of peripheral muscle oxygenation (% SmO2) using near-infrared spectroscopy (NIRS) during exercise in an endurance test during a respiratory rehabilitation session.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric ROCHE, MD-PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Sint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: Undecided